CLINICAL TRIAL: NCT01440270
Title: Neo-adjuvant Erbitux-based Chemotherapy Followed by Surgery and Radiotherapy for Locally Advanced Oral/Oropharyngeal Cancer
Brief Title: Neo-adjuvant Erbitux-based Chemotherapy for Locally Advanced Oral/Oropharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Fudan University (Other); Tongji University (Other); Second Military Medical University (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 622022237
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced Malignant Neoplasm; Oral Cancer; Oropharyngeal Carcinoma
Keywords: Oral cancer; Oropharyngeal cancer; Induction chemotherapy; Targeted chemotherapy; Surgery; Radiotherapy; Effects of Chemotherapy
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neo-adjuvant Erbitux-based chemotherapy (Experimental): Neo-adjuvant Erbitux-based chemotherapy before surgery: Erbitux, Docetaxel, Cisplatin.
  Interventions: Drug: Neo-adjuvant Erbitux-based chemotherapy

INTERVENTIONS:
Drug: Neo-adjuvant Erbitux-based chemotherapy — Name/Substance: Erbitux Formulation: 2 mg/ml or 5 mg/ml Dose: 400 mg/m^2 initial, and then 250 mg/m^2 weekly Route: Intravenous infusion Frequency & treatment mode: Weekly Duration: 6 weeks
  Name/Substance: Docetaxel Formulation: Liquid (20 mg/2 ml) Dose: 75 mg/m^2 Route: Intravenous infusion Frequency & treatment mode: Day 1, every 3 weeks Duration: 2 cycles (6 weeks)
  Name/Substance: Cisplatin Formulation: Powder (30 mg) Dose: 75 mg/m^2 Route: Intravenous infusion Frequency & treatment mode: Day 1, every 3 weeks Duration: 2 cycles (6 weeks)
  Arms: Neo-adjuvant Erbitux-based chemotherapy
  Other Names: Followed by surgery and radiotherapy

SUMMARY:
Epidermal growth factor receptor（EGFR） is a potential target for new anticancer therapy in head and neck squamous cell carcinoma, because blocking the EGFR by a monoclonal antibody results in inhibition of the stimulation of the receptor, therefore, in inhibition of cell proliferation, enhanced apoptosis, and reduced angiogenesis, invasiveness and metastases. The study hypothesis is that neo-adjuvant Erbitux-based chemotherapy followed by surgery and radiotherapy for locally advanced oral/oropharyngeal cancer could benefit the patients on prognosis. The endpoints of this study are the pathological complete response after neo-adjuvant Erbitux-based chemotherapy followed by surgery and radiotherapy, the survival rate, and the safety.

DETAILED DESCRIPTION:
The primary endpoint of this study is the pathological complete response after neo-adjuvant Erbitux-based chemotherapy followed by surgery and radiotherapy. The second endpoint of this study is the disease free survival rates (1, 2, 3, 5 years), locoregional control rates (1, 3, 5 years), overall survival rate (3, 5 years), and the safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study activities
* Age 18-75
* Histological/cytological and iconography confirmed squamous-celled oral/oropharyngeal cancer
* Stage Ⅲ/Ⅳa (T1-2, N1-2, M0 or T3-4, N0-2, M0, AJCC 2010), operable disease
* Karnofsky performance status (KPS) ≥ 70
* Adequate hematologic function: Neutrophils ≥ 1,500/mm^3, WBC > 4,000/mm^3, Hb > 10 g/dL, platelet count > 100,000/mm^3
* Hepatic function: ALAT/ASAT < 2.5 times the upper limit of normal (ULN), bilirubin < 1.5 x ULN
* Renal function: serum creatinine < 1.5 x ULN
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Evidence of distant metastatic disease and other oropharyngeal cancers
* Surgical procedure of the primary tumor or lymph nodes (except diagnostic biopsy) before study treatment
* Previous radiotherapy for the primary tumor or lymph nodes
* Previous exposure to epidermal growth factor - targeted therapy
* Prior chemotherapy or immunotherapy for the primary tumor
* Other previous malignancy within 5 years, except adequately treated non-melanoma skin cancer or pre-invasive carcinoma of the cervix
* Any investigational agent prior to the 1st study medication
* Participation in another clinical study within the 30 days prior to Inclusion in this study.
* Peripheral neuropathy > grade 1
* Known grade 3 or 4 allergic reaction to any of the study treatment
* Creatinine Clearance < 30 ml/min
* Know drug abuse / alcohol abuse
* Legal incapacity or limited legal capacity
* Active systemic infection
* Medical or psychiatric illness, which in the investigators' opinions, would not permit the subject to complete or fully and completely understand the risks and potential complications of the study
* Concurrent chronic systemic immune therapy or hormone therapy not indicated in the study protocol
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period
* Severe cardiac disease such as heart failure, clinically relevant cardiac dysrhythmias, coronary artery disease or myocardial infarction within the last 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response | Up to 6 months
  To evaluate pathological Complete Response (pCR) after neo-adjuvant Erbitux-based chemotherapy followed by surgery and radiotherapy.

SECONDARY OUTCOMES:
Disease Free Survival | 5 years
  Disease Free Survival (DFS) rates (1, 2, 3, 5 years)
Locoregional Control rates | 5 years
  Locoregional Control rates (LCR) (1, 3, 5 years)
Overall Survival | 5 years
  Overall Survival (OS) rate (3, 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-ping Zhang, MD, PhD, Study Chair — Department of Oral and Maxillofacial Surger, Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (7):
- China (7):
  - Eye & Ear Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji University Dongfang Hospital, Shanghai, Shanghai Municipality